CLINICAL TRIAL: NCT02929862
Title: A Phase 1/2A Multicenter, Open-Label Study of LYC-55716 in Adult Subjects With Locally Advanced or Metastatic Cancer
Brief Title: Study of LYC-55716 in Adult Subjects With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYC-55716-1001
Record Dates: First submitted 2016-10-05; First posted 2016-10-11 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2018-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — cintirorgon

ARMS (1):
- Single Agent 55716 (Experimental)
  Interventions: Drug: LYC-55716

INTERVENTIONS:
Drug: LYC-55716 — For Phase 1, increasing doses of oral 55716 given BID for a 28 day cycle. For Phase 2A, the RP2D will be administered to patients for 28 day cycles.

SUMMARY:
This is a Phase 1/2A study designed to evaluate the safety and tolerability of increased repeated doses of LYC-55716 in subjects with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Approximately 30 subjects across approximately 5 United States (US) sites will be enrolled in the Phase 1 portion of the study and approximately 69-84 subjects across approximately 15 US sites will be enrolled in the Phase 2A portion of the study.

The Phase 1 portion of the study will follow a 3 + 3 dose-escalation design to evaluate twice-daily (BID) administration of LYC-55716 for DLTs and to determine the MTD and the RP2D for further assessment in Phase 2A. A treatment cycle will consist of 28 days of treatment and subjects may continue to receive subsequent cycles of therapy as long as they do not have clinically significant progressive disease.

In the Phase 2A portion of the study, 69-84 subjects with locally advanced or metastatic solid tumors considered most likely to be responsive to a RORγ agonist will be enrolled and treated at the MTD or RP2D.

Six cohorts of subjects with advanced cancer will be enrolled. Cohorts 1 to 3 will enroll 14 to 19 subjects per cohort. Tumor types include NSCLC (Cohort 1); gastric, esophageal and G-E junction adenocarcinoma (Cohort 2); and SCCHN (Cohort 3). Cohorts 4 to 6 will enroll up to 9 subjects per cohort. Tumor types include ovarian carcinoma (Cohort 4), renal cell carcinoma (Cohort 5), and urothelial carcinoma (Cohort 6).

Primary Study Objectives

Phase 1

* Evaluate the safety and tolerability of LYC-55716
* Determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D)

Phase 2A

• Determine the objective response rate according to response evaluation criteria in solid tumors (RECIST) v1.1.

Secondary Study Objectives

Phase 1

* Evaluate the activity of LYC-55716 by objective response according to RECIST v1.1.
* Determine the durability of any observed objective response

Phase 2A

* Determine the duration of response
* Determine progression-free survival (PFS) and overall survival (OS)
* Determine suitability of the RP2D for further study
* Characterize the pharmacokinetics (PK) of LYC-55716

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and at least 18 years of age.
* Histological or cytological confirmation of advanced unresectable solid tumors, including those subjects who have progressed on standard anticancer therapy and for whom no further therapy that confers clinical benefit is available.
* Subject has an Eastern Cooperative Oncology Group (ECOG) score of 0 1 or Karnofsky Performance Status Score ≥ 70.
* Subject has a life expectancy of at least 12 weeks.
* Subject has adequate organ function as determined by the following laboratory values:

  * Absolute Neutrophil Count* ≥ 1,500/mm3 (≥ 1.5 x 109/L)
  * Platelets* ≥ 100,000/mm3 (≥ 100 x 109/L)
  * Lymphocytes ≥ 0.5 x 109/L
  * Hemoglobin* > 9.0 g/dL
  * Serum Creatinine or Creatinine Clearance** ≤ 1.5 x ULN, > 50 mL/min
  * Total Serum Bilirubin ≤ 1.5 x ULN (< 3.0 mg/dL if subject has Gilbert's syndrome)
  * Liver Transaminases (ALT/AST) ≤ 2.5 x ULN, ≤ 5.0 x ULN if liver metastases present

    * (* = without ongoing growth factor or transfusion support)
    * (** = calculated by Cockcroft and Gault's formula)
    * (ALT = alanine aminotransferase, AST = aspartate aminotransferase, ULN = upper limit of normal)

Exclusion Criteria:

* Subject has received an investigational drug in the 28 day period before the first dose of study drug (or within 5 half-lives if longer) or is currently participating in another interventional clinical trial.
* Subject has known symptomatic brain metastases or leptomeningeal involvement as assessed by CT scan or MRI. Subjects with stable asymptomatic brain metastases or leptomeningeal disease are eligible if they have not required new treatments for this disease in a 28 day period before the first dose of study drug, and anticonvulsants and steroids have not been administered for a period of 2 weeks prior to the first dose of study drug.
* Subject has not recovered from adverse reactions to prior cancer treatment or procedures (surgery, chemotherapy, immunotherapy, radiation therapy) to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or better.
* Subject has a previous (within 5 years) or current malignancy other than the target cancer with the exception of curatively treated local tumors such as carcinoma in situ of the breast or cervix, basal or squamous cell carcinoma of the skin, or prostate cancer with Gleason Grade < 6 and prostate-specific antigen within normal range.

Modifications to Eligibility Criteria for the following specific tumor types:

Phase 2A will be limited to enrolling the following tumor types:

* NSCLC
* Gastric, Esophageal, and G-E Junction Adenocarcinoma
* SCCHN
* Ovarian Carcinoma
* Renal Cell Carcinoma
* Urothelial Carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-12; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Assess Tumor Activity | 8 weeks
  Evaluated according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Lycera Investigational Site, Huntsville, Alabama
  - Lycera Investigational Site, Sacramento, California
  - Lycera Investigational Site, Washington D.C., District of Columbia
  - Lycera Investigational Site, Sarasota, Florida
  - Lycera Investigational Site, Atlanta, Georgia
  - Lycera Investigational Site, Augusta, Georgia
  - Lycera Investigational Site, Chicago, Illinois
  - Lycera Investigational Site, Saint Cloud, Minnesota
  - Lycera Investigational Site, Omaha, Nebraska
  - Lycera Investigational Site, New York, New York
  - Lycera Investigational Site, Durham, North Carolina
  - Lycera Investigational Site, Oklahoma City, Oklahoma
  - Lycera Investigational Site, Portland, Oregon
  - Lycera Investigational Site, Philadelphia, Pennsylvania
  - Lycera Investigational Site, Greenville, South Carolina
  - Lycera Investigational Site, Nashville, Tennessee
  - Lycera Investigational Site, Dallas, Texas
  - Lycera Investigational Site, San Antonio, Texas
  - Lycera Investigational Site, Charlottesville, Virginia
  - Lycera Investigational Site, Fairfax, Virginia